CLINICAL TRIAL: NCT06004362
Title: Complementary and Integrative Medicine as an Online Intervention in Patients With Post-covid Syndrome - a Randomized-controlled Mixed-methods Trial.
Brief Title: Complementary and Integrative Medicine as an Online Intervention in Patients With Post-covid Syndrome After COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHKOnline
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Post-COVID Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complementary and Integrative Medicine online intervention, routine care and book (Experimental)
  Interventions: Behavioral: Complementary and Integrative Medicine online intervention, routine care and book
- Routine care and book (Active Comparator)
  Interventions: Behavioral: Routine care and book

INTERVENTIONS:
Behavioral: Complementary and Integrative Medicine online intervention, routine care and book — The online program takes place in a multiprofessionally guided online group setting once a week for up to 180 minutes (including several breaks) over a period of 10 weeks:
  * Basic principles of a plant-based whole-food nutrition
  * Procedures of hydrotherapy according to Kneipp
  * Self-help strategies (e.g. teas, wraps, compresses etc.)
  * Methods of mind-body medicine (mindfulness, meditation, breathing, yoga etc.)
  * Methods of extended Complementary and Integrative Medicine (e.g. acupressure)
  It is recommended to practice a part of the taught exercises at home for about 30 minutes daily. In addition, the patients receive a book for the treatment of post-covid syndrome complaints. Group 1 additionally uses the already existing routine care (e.g. general practitioner).
  Arms: Complementary and Integrative Medicine online intervention, routine care and book
Behavioral: Routine care and book — Participants in the second study arm receive routine care, e.g. from their general practitioner. In addition, the patients receive the same book as group 1 for the treatment of post-covid syndrome complaints. The participants of the second study arm will be offered to participate in the Complementary and Integrative Medicine online intervention after 4 months within the study.
  Arms: Routine care and book

SUMMARY:
The Post-COVID syndrome is a COVID-19 sequelae disease with high individual burden. We conduct a prospective, two-arm, randomized-controlled intervention study with embedded qualitative and physiological sub-studies in a mixed-methods design.

ELIGIBILITY:
Inclusion criteria:

* Acute SARS-CoV2 infection at least 12 weeks ago (documented by PCR test results or SARS-CoV-2 antibodies)
* History of chronic fatigue (after SARS-CoV-2 infection)
* At least 3 of 7 criteria fulfilled at the time of inclusion: sleep disturbance, headache, joint pain/muscle pain, anxiety/depression, memory impairment/concentration disturbance, postexertional malaise, dysosmia/anosmia
* Numerical Rating Scale (NRS, 0-10 points, 0 = not able to exercise at all; 10 = full exercise capacity) physical exercise capacity of max. 6 points ("What is your physical exercise capacity on average over the last 7 days?")
* Short Form-36 Physical Function Subscale (SF-36 PFS) of maximum 65 points
* Patient are technically equipped enough to participate in the online intervention and willing to follow the study procedure to perform the online intervention at home

Exclusion criteria:

* Fatigue already present before SARS-CoV-2 infection
* Presence of severe post-exertional malaise (PEM) (according to DSQ-PEM tool question 7 OR 8 with yes AND >14h condition worsening)
* Other underlying conditions leading to symptoms of chronic fatigue, such as unstable mental illness, oncological disease(s), MS, fibromyalgia, and substance abuse
* Other serious underlying medical conditions, such as severe pulmonary, cardiac, psychiatric, or infectious diseases that could interfere with study participation or affect results • Ongoing opioid therapy or opioid therapy in the week prior to study entry
* Regular use of cannabinoids or other illicit drugs in the month prior to or during the study
* Restarting or discontinuing psychotherapy during study participation in the 6 weeks prior to study entry
* Pregnancy or breastfeeding
* Participation in another clinical intervention study during study participation 1
* Regular use of Complementary and Integrative Medicine self-help measures (e.g. meditation, Kneipp hydrotherapiy, etc.) within the study period
* Current pension procedure or planned claiming of a pension procedure due to disability
* Planned rehabilitation measures during study participation due to post-COVID syndrome

Inclusion and exclusion criteria of the sub-study focus group interviews with physicians

Inclusion criteria:

* Family physicians and general practitioners
* Regular outpatient care of patients with post-covid syndrome
* Willingness in principle to participate in a 2-hour interview on-site or online

Exclusion criteria:

• No previous care of post-covid patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Short Form 36 (SF-36), Physical Functioning Scale | Baseline, 10 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.

SECONDARY OUTCOMES:
Short Form 36 (SF-36) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
DePaul Post-Exertional Malaise Questionnaire (DSQ-PEM) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Post-COVID-Syndrom (PCS) Score | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Chalder Fatigue Scale (CFS) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Quality of life (EQ-5D-5L) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
General Self-Efficacy Scale (GSE, German version: ASKU) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Visual analog scale (VAS) physical strength | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Visual analog scale (VAS) mental strength | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Visual analog scale (VAS) headache | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Patient Health Questionnaire 9 (PHQ9) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Lifestyle questions (diet, alcohol, cigarettes, relaxation, hydrotherapie, nature stays, physical activity) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
Expectation regarding study intervention | Baseline
  5-point likert-scale. The scale ranges from 0 to 5, where 0 is the lowest level and 5 is the highest level.
Perceived Stress Scale (PSS 4) | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  The scale ranges from 0 to 100, where 0 is the lowest level and 100 is the highest level.
Satisfaction with the intervention | Week 10
  5-point likert-scale. The scale ranges from 0 to 5, where 0 is the lowest level and 5 is the highest level.
Safety by recording adverse events | Baseline, 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
Adherence to the study intervention | Week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10
  Asking Minutes (min.) of the last week
Online diaries for assessing routine care (GP prescriptions/measures, especially medication and phytotherapy/nutritional supplements) | Week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 20, week 30, week 40, week 50
Continuation of the intervention | 10 weeks, 20 weeks, 30 weeks, 40 weeks, 50 weeks
  Asking Minutes (min.) of the last month

OTHER OUTCOMES:
Qualitative data | Week 10
  After the end of the intervention, qualitative data will be collected at week 10 from a randomized subpopulation (n=15-20) for the purpose of evaluating the online intervention from the patient's perspective using semi-structured, guided interviews with narrative components (of interest, for example, are the subjective experiences, the experience of the disease and its effects).
Sub-study: Focus group interviews with physicians | Week 10
  In a sub-study, focus group interviews will be conducted with n=7-10 primary care physicians in routine care. Depending on the research results, the number and structure of the interviews and the interviewed patients can be adapted according to the explorative requirements of the qualitative analysis. The interviews will be digitally recorded, pseudonymously transcribed and qualitatively analyzed.
Sub-study: biosignal characteristics | Baseline, week 10
  In another subgroup (electrophysiological sub-study) with n=48 participants, multichannel electrophysiological measurements are performed in each case at baseline and week 10, in which heart rate, blood pressure, respiratory rate, pulse, electrodermal activity and brain activity (EEG) are recorded synchronously - by means of monitoring systems (SOMNOmedics, SOMNO HD EEG 32) and Corsano Smartwatch. Furthermore, hand force is measured in a standardized way.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided